CLINICAL TRIAL: NCT02352779
Title: Feasibility of Omega-3 Supplementation for Cancer-Related Fatigue
Brief Title: Omega-3 Fatty Acid in Reducing Cancer-Related Fatigue in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Principal Investigator, URCC NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: URCC13091; NCI-2014-01191 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC13091 (Other: University of Rochester NCORP Research Base); URCC-13091 (Other: DCP); URCC-13091 (Other: CTEP); U10CA037420 (NIH); UG1CA189961 (NIH); R03CA175599 (NIH)
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Breast Carcinoma; Cancer; Fatigue
Keywords: Cancer Survivor
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Fatigue | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (low-dose omega-3 fatty acid) (Experimental): Patients receive low-dose omega-3 fatty acid supplementation PO BID and placebo PO BID for 6 weeks.
  Interventions: Dietary Supplement: Omega-3 Fatty Acid; Other: Placebo; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis
- Arm II (high-dose omega-3 fatty acid) (Experimental): Patients receive high-dose omega-3 fatty acid supplementation PO BID for 6 weeks.
  Interventions: Dietary Supplement: Omega-3 Fatty Acid; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis
- Arm III (placebo) (Placebo Comparator): Patients receive placebo PO BID for 6 weeks.
  Interventions: Other: Placebo; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid — Given PO
  Other Names: O3FA; Omega-3 Fatty Acids; Omega-3 PUFA
  Arms: Arm I (low-dose omega-3 fatty acid); Arm II (high-dose omega-3 fatty acid)
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Arm I (low-dose omega-3 fatty acid); Arm III (placebo)
Other: Questionnaire Administration — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized pilot clinical trial studies omega-3 fatty acid in reducing cancer-related fatigue in breast cancer survivors. Supplementation with omega-3 fatty acid may help reduce cancer-related fatigue in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To collect preliminary statistical data (mean changes and standard deviations) on two omega-3 supplementation (omega-3 fatty acid) regimens (1.65 g/day and 3.3 g/day) compared to placebo for reducing cancer-related fatigue (CRF) in fatigued breast cancer survivors.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive low-dose omega-3 fatty acid supplementation orally (PO) twice daily (BID) and placebo PO BID for 6 weeks.

ARM II: Patients receive high-dose omega-3 fatty acid supplementation PO BID for 6 weeks.

ARM III: Patients receive placebo PO BID for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of breast cancer; participants can have had more than one primary cancer diagnosis in the past
* Have undergone some type or combination of standard adjuvant treatment (surgery, chemotherapy, radiation therapy) for breast cancer
* Have completed all forms of standard adjuvant treatment (surgery, chemotherapy, radiation therapy) for breast cancer between 4 and 36 months prior to enrollment in the study; participants can be currently taking hormones (such as tamoxifen) or monoclonal antibodies (such as Herceptin)
* Must have cancer-related fatigue, as indicated by a response of 4 or greater when asked to rate their level of fatigue at its worst in the past week on an 11-point scale anchored by "0" = no fatigue and "10" = as bad as you can imagine
* Be able to read English
* Able to swallow medication
* Give written informed consent

Exclusion Criteria:

* Have used marine omega-3 supplements at any time within previous 3 months (this includes prescription omega-3 drugs such as Lovaza®)
* Be taking anticoagulant medication (does not include aspirin)
* Have sensitivity or allergy to fish and/or shellfish
* Have sensitivity or allergy to soy and/or soybeans
* Have confirmed diagnosis of chronic fatigue syndrome or other diagnosis known to cause severe fatigue

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke Peppone, Principal Investigator — University of Rochester NCORP Research Base
Locations (6):
- United States (6):
  - Wichita NCORP, Wichita, Kansas
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - University of Rochester NCORP Research Base, Rochester, New York
  - Dayton NCORP, Dayton, Ohio
  - Greenville Health System NCORP, Greenville, South Carolina
  - Wisconsin NCORP, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kleckner AS, Kleckner IR, Culakova E, Wojtovich AP, Klinedinst NJ, Kerns SL, Hardy SJ, Inglis JE, Padula GDA, Mustian KM, Janelsins MC, Dorsey SG, Saligan LN, Peppone LJ. Exploratory Analysis of Associations Between Whole Blood Mitochondrial Gene Expression and Cancer-Related Fatigue Among Breast Cancer Survivors. Nurs Res. 2022 Sep-Oct 01;71(5):411-417. doi: 10.1097/NNR.0000000000000598. Epub 2022 Apr 13. PMID 35416182
- [Derived] Inglis JE, Kleckner AS, Lin PJ, Gilmore NJ, Culakova E, VanderWoude AC, Mustian KM, Fernandez ID, Dunne RF, Deutsch J, Peppone LJ. Excess Body Weight and Cancer-Related Fatigue, Systemic Inflammation, and Serum Lipids in Breast Cancer Survivors. Nutr Cancer. 2021;73(9):1676-1686. doi: 10.1080/01635581.2020.1807574. Epub 2020 Aug 19. PMID 32812824
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/publications/pdq

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Low-dose Omega-3 Fatty Acid) | Arm II (High-dose Omega-3 Fatty Acid) | Arm III (Placebo)
Started | 37 | 36 | 35
Completed | 29 | 35 | 33
Not Completed | 8 | 1 | 2
Not completed — Personal Issues | 1 | 1 | 0
Not completed — Too Many Forms | 2 | 0 | 0
Not completed — Feeling Overwhelmed | 1 | 0 | 0
Not completed — Disliked Intervention | 1 | 0 | 0
Not completed — Changed Mind | 1 | 0 | 0
Not completed — Study Related Symptoms | 1 | 0 | 0
Not completed — Absence of Symptoms | 1 | 0 | 0
Not completed — Other Medical Reason | 0 | 0 | 1
Not completed — No Reason | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Low-dose Omega-3 Fatty Acid) | Arm II (High-dose Omega-3 Fatty Acid) | Arm III (Placebo) | Total
Number analyzed (Participants) | 29 | 35 | 33 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.62 (11.10) | 60.40 (9.35) | 58.03 (10.94) | 59.66 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 33 | 97
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 35 | 33 | 96
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 5
  White | 27 | 31 | 33 | 91
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Values below 18.5 represent "Underweight", 18.5 to 24.9 represent "Normal or Healthy Weight", 25.0 to 29.9 represent "Overweight" and 30.0 and above represent "Obese".
  kg/m^2 | 30.11 (6.07) | 32.31 (7.45) | 32.64 (8.17) | 31.76 (7.34)
Karnofsky Performance Status (KPS) [Mean (Standard Deviation); unit: Karnofsky Performance Scale] — The Karnofsky Performance Scale (KPS) Index allows patients to be classified as to their functional impairment. Essentially as used in oncology, the KPS is a measure of time to death. A higher score is favorable. There are 3 general categories which are broken down into 11 specific criteria. Scale range is from 0 (Dead) to 100 (Normal, no complaints, no evidence of disease). The scale increases in units of 10.
  Karnofsky Performance Scale | 91.38 (5.81) | 92.00 (6.32) | 89.70 (7.70) | 91.03 (6.69)
Education Level [Count of Participants; unit: Participants]
  Graduate Degree | 6 | 5 | 4 | 15
  2 or 4 year Degree / Some college | 13 | 18 | 14 | 45
  HS / GED Degree | 10 | 12 | 14 | 36
  No HS Degree or GED | 0 | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants]
  Married | 16 | 20 | 25 | 61
  Long Term, Committed SO | 2 | 0 | 3 | 5
  Divorced | 5 | 7 | 0 | 12
  Single | 3 | 4 | 2 | 9
  Widowed | 3 | 4 | 3 | 10
Employment Status (Current) [Count of Participants; unit: Participants]
  Employment outside the house | 16 | 18 | 13 | 47
  Self Employed | 3 | 3 | 0 | 6
  Home Maker | 6 | 3 | 9 | 18
  Unemployed | 4 | 11 | 11 | 26
Previous Treatment - Surgery [Count of Participants; unit: Participants]
  Yes | 28 | 33 | 33 | 94
  No | 1 | 2 | 0 | 3
Previous Treatment - Chemotherapy [Count of Participants; unit: Participants]
  Yes | 13 | 19 | 17 | 49
  No | 16 | 16 | 16 | 48
Previous Treatment - Radiation [Count of Participants; unit: Participants]
  Yes | 19 | 28 | 25 | 72
  No | 10 | 7 | 8 | 25
Previous Treatment - Hormone Therapy [Count of Participants; unit: Participants]
  Yes | 2 | 6 | 9 | 17
  No | 27 | 29 | 24 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Change (6 Weeks - Baseline) and Standard Deviation in Cancer-related Fatigue, Using the Brief Fatigue Inventory-Short Form (BFI-SF) and Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF). 81 Subjects Had Both a Baseline and 6 Week Value
Description: BFI-SF is a 4 item questionnaire to assess the severity of fatigue, ranging from 0 (No Fatigue) to 10 (As bad as you can imagine).
  MFSI-SF is a 30 item questionnaire to assess the level of fatigue in terms of general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor). First four subscales (general, physical, emotional, and mental) are summed and the vigor scale is subtracted to create fatigue total score with a range of -32 (low fatigue) to 96 (high fatigue).
Time Frame: Baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Low-dose Omega-3 Fatty Acid) | Arm II (High-dose Omega-3 Fatty Acid) | Arm III (Placebo)
Number analyzed (Participants) | 24 | 30 | 27
units on a scale
  BFI-SF Mean Post - Pre | -3.66 [-4.37 to -2.96] | -3.68 [-4.31 to -3.05] | -2.99 [-3.65 to -2.33]
  MFSI-SF Mean Post - Pre | -11.03 [-16.55 to -5.50] | -13.93 [-18.82 to -9.05] | -10.94 [-16.07 to -5.82]
Statistical Analysis 1: Comparison: Arm I (Low-dose Omega-3 Fatty Acid) vs Arm III (Placebo); BFI-SF; Test type: Other; p = 0.1666, ANCOVA; Based on a contrast using the three-arm ANCOVA; Mean Difference (Final Values) = 0.6763, Standard Error of Mean 0.4843
Statistical Analysis 2: Comparison: Arm II (High-dose Omega-3 Fatty Acid) vs Arm III (Placebo); BFI-SF; Test type: Other; p = 0.1329, ANCOVA; Based on a contrast using the three-arm ANCOVA; Mean Difference (Final Values) = 0.6936, Standard Error of Mean 0.4567
Statistical Analysis 3: Comparison: Arm I (Low-dose Omega-3 Fatty Acid) vs Arm III (Placebo); MFSI-SF; Test type: Other; p = 0.9826, ANCOVA; Based on a contrast using the three-arm ANCOVA; Mean Difference (Final Values) = 0.0831, Standard Error of Mean 3.8065
Statistical Analysis 4: Comparison: Arm II (High-dose Omega-3 Fatty Acid) vs Arm III (Placebo); MFSI-SF; Test type: Other; p = 0.4016, ANCOVA; Based on a contrast using the three-arm ANCOVA; Mean Difference (Final Values) = 2.9898, Standard Error of Mean 3.5448

ADVERSE EVENTS:
Arm/Group | Arm I (Low-dose Omega-3 Fatty Acid) | Arm II (High-dose Omega-3 Fatty Acid) | Arm III (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/29 | 0/35 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low-dose Omega-3 Fatty Acid) (N=29) | Arm II (High-dose Omega-3 Fatty Acid) (N=35) | Arm III (Placebo) (N=33)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No